CLINICAL TRIAL: NCT04571632
Title: A Randomized Phase II Clinical Trial of SBRT and Systemic Pembrolizumab With or Without Intratumoral Avelumab/Ipilimumab Plus CD1c (BDCA-1)+/ CD141 (BDCA-3)+ Myeloid Dendritic Cells in NSCLC Subtitle v3.0: A Randomized Phase II Clinical Trial of SBRT and Systemic Pembrolizumab With or Without Intratumoral Avelumab/Ipilimumab Plus CD1c (BDCA-1)+/CD141 (BDCA-3)+ Myeloid Dendritic Cells in Solid Tumors.
Brief Title: Clinical Trial of SBRT and Systemic Pembrolizumab With or Without Avelumab/Ipilimumab+ Dendritic Cells in Solid Tumors
Acronym: Luscid
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-BN-001
Record Dates: First submitted 2020-09-08; First posted 2020-10-01 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-02

CONDITIONS: Non Small Cell Lung Cancer; Solid Tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Ipilimumab; pembrolizumab; Injections; Antigens, CD1d

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate treatment arm: (Active Comparator): On day -3, -1 and 1, SBRT fractions of 8 Gy will be administered to subjects. On day 1, approximately 2 hours after the last SBRT fraction, intratumoral injection of ipilimumab (Yervoy®, 50mg/10mL solution) at a maximum total dose of 10 mg (= 2 ml of a 50mg/10ml solution) and avelumab (Bavencio®, 200mg/10mL solution) at maximum total dose of 40 mg (= 2 ml of a 200mg/10ml solution) will be performed. Subject will also receive a standard 200mg (fixed dose) intravenous infusion of pembrolizumab (Keytruda®, 100 mg/4mL solution).
  On day 2, autologous, non-substantially manipulated CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC will be intratumorally administered. Previously cryopreserved CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC will be thawed before administration.
  On day 21 and every 21 days thereafter, IT injection of ipilimumab and avelumab and IV pembrolizumab at the same dose as on day 1 will be performed. Treatment will be discontinued upon disease progression
  Interventions: Drug: Avelumab; Drug: Ipilimumab 5 MG/ML; Drug: Pembrolizumab 100 MG in 4 ML Injection; Other: CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC
- Contemporary control arm (Active Comparator): On day -3, -1 and 1, SBRT fractions of 8 Gy will be administered to subjects. On day 1 and every + 21 days thereafter, subjects will receive a standard 200mg (fixed dose) IV pembrolizumab (Keytruda®, 100 mg/4mL solution) dose.
  On disease progression, intratumoral administration as in the "immediate-treatment" arm will be conducted. Thus, intratumoral injection of ipilimumab at a maximum total dose of 10 mg and avelumab at maximum total dose of 40 mg will be performed. Administration of pembrolizumab at a dose of 200 mg will be continued.
  Tumor response assessments by whole body PET/CT will be scheduled in week 12 and every 12 weeks thereafter during the treatment phase; . Baseline scan will be performed during screening period Procurement of tumor tissue by fine needle aspirates will be performed at the time of every intra-tumoral study drug administration
  Interventions: Drug: Avelumab; Drug: Ipilimumab 5 MG/ML; Drug: Pembrolizumab 100 MG in 4 ML Injection; Other: CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC

INTERVENTIONS:
Drug: Avelumab — Avelumab (200mg/10mL solution) will be administered by intratumoral injection at a maximum total dose of 40 mg (= 2 ml of a 200mg/10ml solution) on day 1 followed by a subsequent intratumoral injections on day 15, 29, 43, 57 and 71.
  Total administered dose of avelumab (200mg/10mL solution) will be up to 2.0 mL per treatment. Injected volume per lesion will range from 0.05 mL for lesions < 0,5 cm to 2.0 mL for lesions > 5 cm in longest diameter.
  Injection of all lesions in individual patients will not be required.
  Other Names: Bavencio
Drug: Ipilimumab 5 MG/ML — Ipilimumab (50mg/10mL solution) will be administered by intratumoral injection at a maximum total dose of 10 mg (= 2 ml of a 50mg/10ml solution) on day 1 followed by a subsequent intratumoral injections on day 15, 29, 43, 57 and 71.
  Total administered dose of ipilimumab (50mg/10mL solution) will be up to 2.0 mL per treatment. Injected volume per lesion will range from 0.05 mL for lesions < 0,5 cm to 2.0 mL for lesions > 5 cm in longest diameter.
  Injection of all lesions in individual patients will not be required. Determination of ipilimumab (50mg/10mL solution) injection volume based on lesion size
  Other Names: Yervoy
Drug: Pembrolizumab 100 MG in 4 ML Injection — The first administration of pembrolizumab 200 mg (100 mg/4mL solution) by the intravenous route during 30 minutes will be administered on day 1. The second administrations of pembrolizumab 200 mg will be administered by a 30 minutes intravenous infusion on day 21, and thereafter every 21 days (or up to ± 3 days before or after the scheduled date if necessary) days.
  Other Names: Keytruda
Other: CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC — CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC will be administered by intratumoral injection in the lesions that were injected by avelumab en ipilimumab on day 1 (approximately 24 hours after intratumoral injection of avelumab en ipilimumab).
  The total administered CD1c (BDCA-1)+/ CD141 (BDCA-3)+ myDC volume will be up to 4.0 mL per intratumoral treatment session. Injected volume per lesion (skin-, soft tissue or lymph-node metastases) will range from 0.1 mL for lesions < 0,5 cm to 4.0 mL for lesions > 5 cm in longest diameter. Injection of all lesions in an individual patient will not be required.
  The determination of CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC injection volume is based on lesion size.
  When lesions are clustered together, they are injected as a single lesion according to the table for determination of CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC injection volume based on lesion size.

SUMMARY:
A randomized phase II clinical trial of SBRT and systemic pembrolizumab with or without intratumoral avelumab/ipilimumab plus CD1c (BDCA-1)+/CD141 (BDCA-3)+ myeloid dendritic cells in solid tumors.

DETAILED DESCRIPTION:
Cancer cells can be recognized by the patient's own immune system, a process that is referred to as the "cancer immunity cycle" (Chen & Mellman 2013; Mellman 2013; Chen & Mellman 2017).

Remarkable anti-tumor activity has been achieved by blocking the inhibitory T-cell receptor CTLA-4 and/or the PD-1/-L1 axis. Immune checkpoint inhibition by monoclonal antibody (mAb) therapy has become a standard of care in patients with advanced melanoma, renal cell carcinoma, non-small cell lung carcinoma, Hodgkin's lymphoma and bladder cancer. Indications are continuously expanding. Activity of PD-1/-L1 and CTLA-4 inhibition has been correlated with hallmarks of pre-existing anti-tumor T-cell response (presence of activated cytotoxic T lymphocytes (CTL) in the tumor microenvironment (TME) as evident from transcription profiles) and PD-L1 expression by tumor cells (in response to T-cell secreted IFN-). Mutational load of the cancer cells and presence of highly immunogenic neo-epitopes in the cancer cell genome underlies the capacity for cancer cells to elicit an immune response (Tumeh, Harview et al. 2014). Responsiveness to treatment with CTLA-4 has been correlated with the expression of HLA class I molecules by the cancer cells (Tumeh, Harview et al. 2014).

In immune-evasive tumors a pivotal role has been attributed to the elimination of myeloid dendritic cells (myDC) from the TME. myDC play a pivotal role in the initiation and coordination of the activity of anti-tumor CTL activity within the TME (Rodig, Gusenleitner et al. 2017). In animal models, myDC have been demonstrated to play an essential role in "licensing" anti-tumor CTLs to eradicate tumor cells. Activation of oncogenic signaling pathways such as the WNT/Catenin pathway can lead to the exclusion of myeloid DC from the TME (Broz et al. 2014; Spranger & Gajewski 2016). Absence of myDCs at the invasive margin and within metastases has been correlated with defective CTL activation allowing the metastasis to escape the anti-tumor immune response (Salmon, Idoyaga et al. 2016). These myDC also migrate to tumor-draining lymph nodes and present tumor antigens to T-cells in these secondary lymphoid organs (Salmon, Idoyaga et al. 2016). In mouse models, tumor-residing Batf3 dendritic cells were shown to be required for effector T Cell trafficking and success of adoptive T-cell therapy (Roberts et al. 2016). Presence of myeloid DC's was more strongly correlated with a "T-cell inflamed TME signature" as compared to neo-antigen load in 266 melanomas from The Cancer Genome Atlas (Spranger, Luke et al. 2016).

Two important human myDCs subsets exist that are differentiated by expression of either the BDCA-1 or BDCA-3 surface marker. The CD1c (BDCA-1)+ antigen is specifically expressed on human dendritic cells, which are CD11chighCD123low and represent the major subset of myDCs in human blood (about 0.6 % of all peripheral blood mononuclear cells (PBMCs)). CD1c (BDCA-1)+ myDC have a monocytoid morphology and express myeloid markers such as CD13 and CD33 as well as Fc receptors such as CD32, CD64, and FceRI. Furthermore, myDC are determined to be CD4+, Lin (CD3, CD16, CD19, CD20, CD56)-, CD2+, CD45RO+, CD141 (BDCA-3)-, CD303 (BDCA-2)-, and CD304 (BDCA-4/Neuropilin-1)-.

A proportion of CD1c (BDCA-1)+ myDC co-expresses CD14 and CD11b. These dual positive cells for CD14 and CD1c (BDCA-1) have immunosuppressive capacity and inhibit T-cell proliferation in vitro. Depletion of this cell type is preferred prior to using CD1c (BDCA-1)+ cells for immune-stimulatory purposes (Bakdash, Buschow et al. 2016).

CD1c (BDCA-1)+ myDC play an important role in the cross-presentation of tumor antigens following immunogenic cell death (Di Blasio, Wortel et al. 2016). Under conditions of tumor growth, myDC will be poorly recruited to the tumor microenvironment, do not get activated and thereby fail to efficiently coordinate anti-tumor immunity within the tumor micro-environment and present tumor associated antigens within tumor-draining lymph nodes. When activated appropriately, human CD1c (BDCA-1)+ dendritic cells secrete high levels of IL-12 and potently prime CTL responses (Di Blasio, Wortel et al. 2016). In vitro, IL-12 production by CD1c (BDCA-1)+ myDC can be boosted by exogenous IFN-(Nizzoli, Krietsch et al. 2013) CD1c (BDCA-1)+ myDC spontaneously "partially mature" within 12 hours following their isolation. Optimal maturation with secretion of IFN- as well as the orientation of stimulated T-lymphocytes towards a Th1 phenotype is only achieved following Toll-like receptor stimulation (Nizzoli, Krietsch et al. 2013).

Animal models have established the safety and efficacy of intra-tumoral administration of ipilimumab. An intratumoral dose of CTLA-4 blocking mAb administered at a ratio of [1:100] compared to intravenous dosing was found to result in equivalent anti-tumor effect and was associated with less systemic toxicity (Skold, van Beek et al. 2015) (Marabelle, Kohrt et al. 2013). In an ongoing clinical trial for patients with advanced melanoma, conducted by our research group, intratumoral injection of CD1c (BDCA-1)+ myDC together with the CTLA-4 blocking mAb ipilimumab plus intravenous administration of the PD-1 blocking mAb nivolumab have been proven feasible and safe. Intratumoral administration of an anti-PD-L1 IgG1 mAb may increase the potential for antibody dependent cellular cytotoxicity (ADCC) and complement dependent cytotoxicity (CDC).

Additionally, the investigators have previously investigated the utility of SBRT to primary tumor and metastatic locations in oligometastatic non-small cell lung carcinoma (NSCLC) patients and found that this treatment was feasible, safe and resulted in an overall metabolic response rate in 60% of the treated population, with 30% of patients achieving a complete metabolic remission (Collen, Christian et al. 2014). Radiation therapy (RT) has been recognized as potentially synergistic with immune checkpoint blockade. Tumor cell killing by radiation results in release of tumor antigens, reduces the immunosuppression within the TME and can reinvigorate the cancer-immunity cycle by upregulation of immunogenic cell surface markers and inducing immunogenic cell death (Dewan, Galloway et al. 2009; Kulzer, Rubner et al. 2014; Frey, Ruckert et al. 2017). Moreover, it has been shown that RT-induced immunogenic cell death can trigger DC maturation and activation in vitro (Kulzer et al. 2014), providing a clear rationale for combining DC-therapy together with RT.

In this randomized phase II clinical trial, the investigators propose to conduct hypofractionated SBRT in combination with systemic PD-1 immune checkpoint blockade (pembrolizumab) with or without intratumoral PD-L1/CTLA-4 inhibition plus intratumoral administration of CD1c (BDCA-1)+ / CD141 (BDCA-3)+ myDC.

ELIGIBILITY:
Inclusion Criteria:

* • Subject has provided written informed consent prior to initiation of any study-specific activities/procedures.

  * Male or female age ≥ 18 years at the time of informed consent.
  * All subjects must have histologically confirmed advanced solid tumors that cannot be completely surgically resected All subjects must have received prior pembrolizumab or nivolumab (with or without cytotoxic chemotherapy or other additional drugs) and fail to respond to this treatment (patients must be documented with stable or progression of disease as their best response to this first-line therapy).
  * Oligometastatic" disease defined by a number of metastatic sites 7
  * ECOG performance status of 0 or 1
  * Patients need to have ≥ 1 metastatic lesion (≥ 10 mm in longest diameter) that can be safely injected by ultrasound-/ CT-guidance, by endo-bronchial ultrasound (EBUS) or even clinically. The lesion should also be amenable for safe biopsy.
  * Injectable metastasis need(s) to be eligible for SBRT
  * Adequate organ function determined within 14 days prior to enrollment
  * Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  * Subject has a tumor sample (a representative archival tissue sample obtained prior to study participation or newly obtained biopsy). Subject must submit the tumor sample during screening. Subjects with a nonevaluable archival sample may obtain a new biopsy and subjects with a non-evaluable newly obtained biopsy may undergo re-biopsy at the discretion of the investigator.
  * Subjects should have adequate vascular access to undergo a leukapheresis

Exclusion Criteria:

* Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids >8 mg/day of methylprednisone or equivalent. The exception does not include leptomeningeal metastasis which is excluded regardless of clinical condition.

  * History or evidence of active autoimmune disease that requires systemic treatment Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * History or evidence of immunodeficiency states (eg, hereditary immune deficiency, organ transplant, or leukemia)
  * History of serious immune related adverse event during treatment with pembrolizumab in first-line
  * History of other malignancy within the past 5 years of enrollment Prior treatment with immune-checkpoint inhibitors (including but not restricted to PD-1, PD-L1 and CTLA-4 blocking mAb) biological cancer therapy, targeted therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment. Subjects should not have ongoing grade 3 or 4 immune-related or chemotherapy-related adverse events. Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study Expected to require other cancer therapy while on study with the exception of local radiation treatment to the site of bone and other metastasis for palliative pain management
  * Other investigational procedures while participating in this study are excluded.
  * History or evidence of symptomatic autoimmune pneumonitis, glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, or active autoimmune disease or syndrome that has required systemic treatment in the past 2 years
  * Evidence of clinically significant immunosuppression
  * Known human immunodeficiency virus (HIV) disease
  * Known acute or chronic hepatitis B or hepatitis C infection
  * Known syphilis infection
  * Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 6 months after the last dose of study treatment
  * Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 6 months after the last dose of study treatment Postmenopausal (therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.) Male subject who is unwilling to use acceptable method of effective contraception during trial participation and through 6 months after the last dose of study treatment. For this trial, male subjects will be considered to be of non-reproductive potential if they have azoospermia (whether due to having had a vasectomy or due to an underlying medical condition). Note: Acceptable methods of effective contraception are defined in the informed consent form.
  * Subject has known sensitivity to any of the products or components to be administered during dosing.
  * Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge
  * History or evidence of psychiatric, substance abuse, or any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
  * Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or sponsor staff directly involved in this trial, unless prospective institutional review board (IRB)/independent ethics committee (IEC) approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
  * Sexually active subject who is unwilling to use a barrier method (male or female condom) to avoid potential study drug transmission during sexual contact during and within 6 months after study treatment.
  * Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Subjects who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of Graft versus Host Disease.)
  * Has a known history of active tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
1 year progression free survival | 1 year
  1 year progression free survival

SECONDARY OUTCOMES:
Adverse events | up to 3 years
  Adverse events from date of study start until the date of first documented progression or date of death from any cause, whichever comes first

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - Uz Brussel, Brussels

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vounckx M, Tijtgat J, Stevens L, Dirven I, Ilsen B, Vandenbroucke F, Raeymaeckers S, Vekens K, Forsyth R, Geeraerts X, Van Riet I, Schwarze JK, Tuyaerts S, Decoster L, De Ridder M, Dufait I, Neyns B. A randomized phase II clinical trial of stereotactic body radiation therapy (SBRT) and systemic pembrolizumab with or without intratumoral avelumab/ipilimumab plus CD1c (BDCA-1)+/CD141 (BDCA-3)+ myeloid dendritic cells in solid tumors. Cancer Immunol Immunother. 2024 Jul 2;73(9):167. doi: 10.1007/s00262-024-03751-0. PMID 38954010